CLINICAL TRIAL: NCT02037906
Title: Comparison of Escalating, Constant and Reduction Energy Output in SWL for Renal Stones: Multi-arm Prospective Randomized Study.
Brief Title: Escalating, Constant and Reduction Energy Output in SWL for Renal Stones
Acronym: SWL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Princess Al-Johara Al-Ibrahim Cancer Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 13/3948/IRB; 13/3948/IRB (Registry Identifier: Institutional Review Board)
Record Dates: First submitted 2014-01-06; First posted 2014-01-16 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2014-01

CONDITIONS: Renal Stones
Keywords: Renal stones; SWL
MeSH Terms: conditions — Nephrolithiasis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Escalating Energy SWL (Experimental): 50 Patients
  Interventions: Radiation: Escalating Energy SWL
- Constant Energy SWL (Experimental): 50 Patients
  Interventions: Radiation: Constant Energy SWL
- Reduction Energy SWL (Experimental): 50 Patients
  Interventions: Radiation: Reduction Energy SWL

INTERVENTIONS:
Radiation: Escalating Energy SWL — Dose escalation, 1500 SW at 18 kv, followed by 1500 SW at 20 kv and the following 1500 SW at 22 kv.
  Arms: Escalating Energy SWL
Radiation: Constant Energy SWL — Constant dose at 20 kv
  Arms: Constant Energy SWL
Radiation: Reduction Energy SWL — Dose reduction, 1500 SW at 22 kv, followed by 1500 SW at 20 kv and the following at 18 kv.
  Arms: Reduction Energy SWL

SUMMARY:
Research Problem: Shock wave lithotripsy (SWL) dramatically changed the management of renal and ureteral calculus disease. In vitro studies suggest that progressive increase in lithotripter energy output voltage could produce the best overall stone comminution in comparison with constant or deescalating energy output. However, it is possible that the beneficial impact of slow rate SWL on comminution of stones and stone free rates has masked any marginal benefits for energy output escalation. The Escalating SW method adds the benefit of less renal tissue injury.

Research Significance:The present study will signifies and evaluates the stone free rates of three groups of patients with renal stones treated with different SWL energy outputs (Escalating, Constant and Reduction energy output).

Research Objectives: The aim of this research project is to study the effect of dose adjustment strategies on success rate of Shock Wave Lithotripsy in the clinical setting and to optimize the conditions for successful Shock Wave Lithotripsy.

Research Methodology: This clinical trial will be conducted at a tertiary care university hospital. 150 patients referred to the Shock wave lithotripsy unit will be evaluated for eligibility to be randomized into three groups (Dose Escalation, Dose reduction and constant dose). Parameter of the three groups will be compared to detect the treatment difference.

DETAILED DESCRIPTION:
Escalating SW amplitude treatment protocols have been shown to be safe on long-term with less harm to kidney tissue. This clinical trial will be conducted at a tertiary care university hospital. All patients referred to the SWL unit will be evaluated for eligibility to be randomized. Randomization process "complete" or "unrestricted" randomization was used to allocate patients to the three arms of the clinical trial where one patient was randomly assigned to one of the three arms blindly.

ELIGIBILITY:
Inclusion Criteria:

* Single stone
* Radio opaque
* Less than 2cm in size
* Renal stone

Exclusion Criteria:

* bleeding disorder,
* urinary tract infection (UTI)
* distal ureteric obstruction

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2014-01; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Stone clearance after escalating shockwave lithotripsy | 14 days after escalating shockwave lithotripsy
  All patients undergo for imaging investigation of the kidneys, ureters, or bladder (KUB) plain x-ray film at day 14 to assess stone free rate. Stone free was defined as no stones or painless fragments less than 4mm. In additions all patients received pre and post shockwave lithotripsy renal ultrasound on day 1 prior and day 1 shockwave lithotripsy to evaluate for shockwave lithotripsy related hematoma formation.

SECONDARY OUTCOMES:
Stone clearance after constant shockwave lithotripsy | 14 days after constant shockwave lithotripsy
  All patients undergo for imaging investigation of the kidneys, ureters, or bladder (KUB) plain x-ray film at day 14 to assess stone free rate. Stone free was defined as no stones or painless fragments less than 4mm. In additions all patients received pre and post shockwave lithotripsy renal ultrasound on day 1 prior and day 1 shockwave lithotripsy to evaluate for shockwave lithotripsy related hematoma formation.

OTHER OUTCOMES:
Stone clearance after reduction shockwave lithotripsy | 14 days after reduction shockwave lithotripsy
  All patients undergo for imaging investigation of the kidneys, ureters, or bladder (KUB) plain x-ray film at day 14 to assess stone free rate. Stone free was defined as no stones or painless fragments less than 4mm. In additions all patients received pre and post shockwave lithotripsy renal ultrasound on day 1 prior and day 1 shockwave lithotripsy to evaluate for shockwave lithotripsy related hematoma formation.

CONTACTS AND LOCATIONS:
Overall Officials: Danny M Rabah, Professor, Principal Investigator — College Of Medicine, King Saud University
Locations (1):
- King Khalid University Hospital, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
Results will be published in per-reviewed journal